CLINICAL TRIAL: NCT04372043
Title: Evaluation of the Sleep Hygiene in the Lebanese Population During the COVID-19 Confinement Period.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Other Study IDs: CEHDF1650
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Sleep Hygiene
MeSH Terms: conditions — Sleep Hygiene | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lebanese population: The "Sleep Hygiene Index" with other demographic questions will be applied to the Lebanese population.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — "Sleep Hygiene Index" and demographic questions.

SUMMARY:
The term "sleep hygiene" refers to a series of healthy sleep habits that can improve the ability to fall asleep. These habits are the most effective long-term treatment for people with chronic insomnia. The "Sleep Hygiene Index" is a 13-item questionnaire that evaluates these habits. We are in the process of validation of this questionnaire in the arabic language.

We will evaluate these habits in the Lebanese population during the COVID-19 confinement period.

DETAILED DESCRIPTION:
The sleep hygiene will be evaluated during the COVID-19 confinement period. The "Sleep Hygiene Index" with other questions will be applied to the Lebanese population in english and arabic. It will be distributed by the means of WhatsApp and Facebook.

ELIGIBILITY:
Inclusion Criteria:

* Lebanese living in Lebanon, 18 YO and over, understanding written english or arabic.

Exclusion Criteria:

* Not having the inclusion criteria.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Lebanese population living in Lebanon during the confinement period of the COVID-19 pandemic.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-04-30 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Sleep Hygiene | 30/04/2020 to 30/12/2020

CONTACTS AND LOCATIONS:
Overall Officials: Jeanine El Helou, MD, MSc, Study Chair — USJ
Locations (1):
- Saint Joseph University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided
Will check with the USJ board